CLINICAL TRIAL: NCT07044596
Title: Non-invasive Stimulation of the Glymphatic System for Slowing Cognitive Decline
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Neuraworx Medical Technologies (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0970; A535700 (Other: UW Madison); Protocol Version 3/10/25 (Other: UW Madison); SMPH/NEURO SURG/NEURO SURG (Other: UW Madison)
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-07

CONDITIONS: Mild Traumatic Brain Injury; Post Concussion Syndrome
MeSH Terms: conditions — Brain Concussion; Post-Concussion Syndrome | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Healthy Controls (Active Comparator)
  Interventions: Device: Functional near-infrared spectroscopy (fNIRS); Device: V1 stimulation electrodes; Device: Magnetic Resonance Imaging (MRI)
- Mild traumatic brain injury (mTBI) (Active Comparator): Participants with recent mTBI
  Interventions: Device: Functional near-infrared spectroscopy (fNIRS); Device: V1 stimulation electrodes; Device: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Device: Functional near-infrared spectroscopy (fNIRS) — fNIRS is a non-invasive imaging technique which takes advantage of the light scattering and absorption differences between oxygenated (HbO) and de-oxygenated hemoglobin (HbDO) to characterize changes in cerebral hemodynamics in response to a given task or stimulus.
Device: V1 stimulation electrodes — The V1 electrodes will be placed on the forehead with some gel and held in place with a headband or cap (a conductive adhesive gel may be placed under the electrodes to help with stimulation). Participants will receive short electrical stimulations through these electrodes that will differ in intensity.
Device: Magnetic Resonance Imaging (MRI) — Participants will undergo 2 90-minute MRI sessions

SUMMARY:
The purpose of this research is to demonstrate that mild stimulation of a nerve (trigeminal nerve) in the head can modulate blood flow in the brain. The modulated blood flow will restore the flow of cerebrospinal fluid (CSF) and this in turn can help improve waste clearance in the brain and prevent build up that may lead to disease.

DETAILED DESCRIPTION:
The goal of this clinical trial is to demonstrate that non-invasive stimulation of the trigeminal nerve can be used to restore blood flow and consequently modulate CSF flow into the brain parenchyma to facilitate brain waste clearance that is impaired in patients with AD. This study will collect brain MRI data on 20 healthy cognitively unimpaired adults receiving intermittent trigeminal nerve branch (V1) mouth stimulation. Participants with recent mild traumatic brain injuries will also be enrolled to establish feasibility within a clinically relevant population.

ELIGIBILITY:
Inclusion Criteria - Healthy Participants :

* Age 20-85 years
* Willing and able to undergo all procedures
* Free of any neurological (e.g., epilepsy, stroke, Parkinson's, brain tumors, moderate or severe traumatic brain injury), neuropsychiatric (e.g., schizophrenia, substance abuse, clinical depression), or developmental (e.g., autism, ADHD) or any other medical condition at the discretion of the PI and co-investigators

Inclusion Criteria - mTBI :

* Age 20-65
* Diagnosed with mild traumatic brain injury and be within 1-52 weeks post-injury
* Willing and able to undergo all procedures

Exclusion Criteria - Healthy Participants:

* Contraindication to MRI
* Known allergies to common electrode materials

Exclusion Criteria - mTBI:

* Contraindications for MRI
* Known allergies to common electrode materials
* Candidates currently on cardiovascular medications which, in the opinion of the investigators, would introduce a confounding factor to glymphatic system function (i.e. ACE-inhibitors, angiotensin receptor blockers, calcium channel blockers)
* Candidates who have chronic infectious diseases (e.g. hepatitis, HIV, TB)
* Candidates diagnosed with small vessel disease, vascular associated dementia (e.g. VCID), or renal disease
* Candidates retinopathies or neuropathies that, in the opinion of the investigators, would prevent them from being able to complete the study or would introduce a confounding factor to glymphatic system function
* Candidates with neurological disorders other than those attributed to their primary diagnosis (e.g. MS, PD, ALS, AD or other dementia, uncontrolled pain)
* Candidates who have had a penetrating injury, craniotomy (with the exception of a burr hole (trephination) for resolution of acute subdural hematoma), or refractory subdural hematoma
* Candidates with a history of seizures (except those in the acute or post-acute phases and are controlled)
* Candidates who experienced a loss of consciousness greater than 24 hours as a result of their TBI
* Candidates who, in the opinion of the investigators, are unable to feel a sensory referred sensation from the stimulation or successfully complete the electrode placement and testing fNIRs

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in blood flow through the brain parenchyma - fNIRS | Baseline to 4 hours
  The fNIRS device will record changes in the blood oxygen level in the brain that is caused by the V1 stimulation.
Change in blood flow through the brain - MRI | Baseline to 90 minutes
  The MRI will record changes in the blood oxygen level in the brain that is caused by the V1 stimulation.
Change in cerebrospinal fluid flow | Baseline to 90 minutes
  MRI scan will be used to measure the flow of cerebrospinal fluid before, during and after stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Kip Ludwig, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No